CLINICAL TRIAL: NCT05833997
Title: Safety Analysis and Oncological Outcomes in Endoscopic Bladder Tumor Resection With Laser Holmium Compared With Transurethral Resection: a Prospective and Randomized Study
Brief Title: Safety Analysis and Oncological Outcomes in HoLERT vs TURBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Alexandre Iscaife, Md, PhD, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP1537/2019
Record Dates: First submitted 2023-04-05; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Bladder Urothelial Carcinoma; Bladder Cancer
Keywords: Bladder urothelial cancer; bladder cancer; transurethral resection of bladder tumor; En-bloc Resection of Bladder Tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium Laser En-bloc Resection of Bladder Tumors (HoLERBT) arm (Experimental): Patients randomized to HoLERBT group will have their tumor resected using the Megapulse 70w (Richard Wolf).
  Interventions: Procedure: Holmium Laser resection of bladder tumor (HoLEBT)
- Control arm (Active Comparator): Patients randomized to control arm will undergo a monopolar transurethral resection of bladder tumor.
  Interventions: Procedure: Monopolar Transurethral resection of bladder tumor

INTERVENTIONS:
Procedure: Monopolar Transurethral resection of bladder tumor — Patients randomized to Monopolar TURBT will be operated using a 26F continuous-flow resectoscope sheaths and a single-pole working element to exclusive use of the resection. The power will be set to cut in 80w and 60w. The technique that will be performed will be the classic endoscopic resection from the top of the tumor until reaching the base, taking a sample from the base of the lesion (muscle layer). Fragments will be removed through an Ellik evacuator, and the solution used will be 3% glycine. After the procedure, the patient will will be catheterized with a silicon catheter number 22F with three ways and continuous irrigation.
  After 30-60 days of the first procedure, all patients diagnosed with a lamina propria invasion in the uro-pathology analysis (T1) will be submitted to a new monopolar TURBT.
  Arms: Control arm
Procedure: Holmium Laser resection of bladder tumor (HoLEBT) — It will be used a 24-26F continuous-flow resectoscope sheath with a specific working element to use with a 600µm fiber to Laser Holmium.
  Patients will be operated with the Megapulse 70w (Richard Wolf) and laser will be set to deliver the energy of 0,5J and 30-40Hz frequency, 15-20W of final energy. The solution used will be 0,9% saline solution. The resection will start from the base of the lesion, reaching the muscle layer to obtain a sample and resection of the whole tumor, without fragmentation. After this, the morcellation will be performed in the apex of tumor sparing the base with a long nephroscope, and the patient will will be catheterized with a silicon catheter number 22F with three ways and continuous irrigation. The morcellated product will be sent to the pathology lab for detailed analysis.
  Arms: Holmium Laser En-bloc Resection of Bladder Tumors (HoLERBT) arm

SUMMARY:
Bladder urothelial cancer is the second most common urologic tumor and represents a worldwide public health problem. Most cases are diagnosed as non-muscle invasive tumors, and can be treated with transurethral resection of bladder tumor (TURBT). However, the electrical energy-based TURBT fragments the tumor, burning it to its own muscular layer leading to artifacts that may spoil the histopathological analysis, resulting in understaging after the first TURBT ranging from 30-64%, depending on the presence of detrusor muscle. Modern laser technologies have been emerging as an alternative to classical TURB using en bloc tumor resection technique (ERBT). Therefore, the laser is applied on tumor's pedicle to resect the whole and intact tumor without fragmentation or fulguration as occurs in TURBT. The purpose of using laser if to improve the resection quality, decrease intra and perioperative complications, avoid re-TURBT and reduce recurrence rates at the resection site and in distant sites. Thus, the purpose of this study is to evaluate Laser Holmium use for large tumors resection (>3cm), reducing complications, costs, and the need for new approaches, and improving the muscle layers samples.

DETAILED DESCRIPTION:
This is a single-institution, randomized, single-blinded, prospective, controlled study, with 2 groups - 50 patients in Holmium Laser En-bloc Resection of Bladder Tumors (HoLERBT) arm and 50 patients in TURBT arm. All the patients will undergo a new procedure between 30-60 days after the first one (monopolar re-TURBT). The laser group will be operated by an experienced surgeon with more than 50 cases of prostate resection. The monopolar TURBT group will be operated by institutions´s surgeons assistants, urologists with more than 2 years of experience in the area and more than 50 surgeries performed. Pathological samples will be analyzed in the FMUSP Urology Laboratory by a pathologist with huge experience in analysis of bladder tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years old;
* Presence of bladder tumor > 3cm without signals of MIBC or advanced disease (US, CT scan or MRI 3 months before surgery)
* Able to understand and willing to sign a written informed consent document
* Satisfactory clinical pre operatory conditions for surgery with regional or general anesthesia.

Exclusion Criteria:

* Previous diagnosis of muscle-invasive bladder cancer;
* Tumor's Invasive aspect (T2 or more) on image (US, TC or RNM);
* Previous TURBT in the last 5 years;
* Urethral stenosis;
* Previous intra-vesical os systemic chemotherapy or radiotherapy;
* Previous treatment with intravesical BCG
* No clinical conditions for regional or general anesthesia;
* Any other significant disease or disorder which, in the opinion of the investigator may either put the participant at risk because of trial participation or may influence the trial result, or the participant's ability ti participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Presence of Detrusor Muscle (DM) on histopathological analysis of morcellated tumor from HoLERBT and TRUBT | Up to 1 month after the first surgery
  Evaluate the presence of muscle layer in the samples of tumor resection

SECONDARY OUTCOMES:
Compare intraoperative an peri-operative complications | During surgery
  Evaluate intra and peri-operative complications (according to Clavien-Dindo scale) between the two groups
Clinical recurrence-free survival | Until 2 years after surgery
  Clinical recurrence-free survival at 3, 6, 9, 12, 15, 18 and 24 months follow-up (US, CT-scan, MRI, cystoscopy, TURBT)
Clinical progression-free survival | Until 2 years of surgery
  Clinical progression-free survival at 3, 6, 9, 12, 15, 18 and 24 months follow-up (US, CT-scan, MRI, TURBT)
Overall and cancer-specific survival | Until 2 years of surgery
  Overall and cancer-specific survival at 13, 6, 9, 12, 15, 18 and 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: William Nahas, MD, PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo (ICESP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Miladi M, Peyromaure M, Zerbib M, Saighi D, Debre B. The value of a second transurethral resection in evaluating patients with bladder tumours. Eur Urol. 2003 Mar;43(3):241-5. doi: 10.1016/s0302-2838(03)00040-x. PMID 12600426
- [Background] Sievert KD, Amend B, Nagele U, Schilling D, Bedke J, Horstmann M, Hennenlotter J, Kruck S, Stenzl A. Economic aspects of bladder cancer: what are the benefits and costs? World J Urol. 2009 Jun;27(3):295-300. doi: 10.1007/s00345-009-0395-z. Epub 2009 Mar 7. PMID 19271220
- [Background] Svatek RS, Hollenbeck BK, Holmang S, Lee R, Kim SP, Stenzl A, Lotan Y. The economics of bladder cancer: costs and considerations of caring for this disease. Eur Urol. 2014 Aug;66(2):253-62. doi: 10.1016/j.eururo.2014.01.006. Epub 2014 Jan 21. PMID 24472711
- [Background] Rink M, Babjuk M, Catto JW, Jichlinski P, Shariat SF, Stenzl A, Stepp H, Zaak D, Witjes JA. Hexyl aminolevulinate-guided fluorescence cystoscopy in the diagnosis and follow-up of patients with non-muscle-invasive bladder cancer: a critical review of the current literature. Eur Urol. 2013 Oct;64(4):624-38. doi: 10.1016/j.eururo.2013.07.007. Epub 2013 Jul 19. PMID 23906669
- [Background] Herrmann TR, Liatsikos EN, Nagele U, Traxer O, Merseburger AS; EAU Guidelines Panel on Lasers, Technologies. EAU guidelines on laser technologies. Eur Urol. 2012 Apr;61(4):783-95. doi: 10.1016/j.eururo.2012.01.010. Epub 2012 Jan 17. PMID 22285403
- [Background] Kramer MW, Rassweiler JJ, Klein J, Martov A, Baykov N, Lusuardi L, Janetschek G, Hurle R, Wolters M, Abbas M, von Klot CA, Leitenberger A, Riedl M, Nagele U, Merseburger AS, Kuczyk MA, Babjuk M, Herrmann TR. En bloc resection of urothelium carcinoma of the bladder (EBRUC): a European multicenter study to compare safety, efficacy, and outcome of laser and electrical en bloc transurethral resection of bladder tumor. World J Urol. 2015 Dec;33(12):1937-43. doi: 10.1007/s00345-015-1568-6. Epub 2015 Apr 25. PMID 25910478
- [Background] Kramer MW, Wolters M, Cash H, Jutzi S, Imkamp F, Kuczyk MA, Merseburger AS, Herrmann TR. Current evidence of transurethral Ho:YAG and Tm:YAG treatment of bladder cancer: update 2014. World J Urol. 2015 Apr;33(4):571-9. doi: 10.1007/s00345-014-1337-y. Epub 2014 Jun 17. PMID 24935098
- [Background] De Nunzio C, Franco G, Cindolo L, Autorino R, Cicione A, Perdona S, Falsaperla M, Gacci M, Leonardo C, Damiano R, De Sio M, Tubaro A. Transuretral resection of the bladder (TURB): analysis of complications using a modified Clavien system in an Italian real life cohort. Eur J Surg Oncol. 2014 Jan;40(1):90-5. doi: 10.1016/j.ejso.2013.11.003. Epub 2013 Nov 12. PMID 24284200